CLINICAL TRIAL: NCT06797596
Title: Clinical Correlation Evaluation of the LIVERFAStTM Test for Diagnosing Important Liver Lesions of Fibrosis and Steatosis Against MR-based Liver Assessment, Magnetic Resonance Elastography (MRE) for Liver Fibrosis and MR-based Assessment of Steatosis, in Adult US Population.
Brief Title: Clinical Correlation Evaluation of the LIVERFASt Test for Diagnosing Important Liver Lesions of Fibrosis and Steatosis Against Magnetic Resonance Elastography (MRE) for Liver Fibrosis and MR-based Assessment of Steatosis, in Adult US Population.
Acronym: LFMRECT
Status: Not yet recruiting | Type: Observational
Sponsor: Fibronostics USA, Inc (Other)
Responsible Party: Sponsor
Other Study IDs: FIBRO-LFASt-MRE-009-2024
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Liver Fibrosis Due to NASH; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Alcohol Liver Disease
Keywords: LIVERFASt; LIVERFASt Test; Noninvasive Test for the Liver; LIVERFASt for MASLD; LIVERFASt for MASH; Fibronostics; Liverfast fibrosis test; Liverfast steatosis test; Liverfast for MASLD and MASH; Liverfast for liver fibrosis; Liverfast plus MRE; Liverfast and MRE; Liverfast and other imaging tools

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective cross-sectional research intended to explore the utility of LIVERFASt in the clinical pathways for the detection of liver fibrosis and steatosis in comparison with the Magnetic Resonance Elastography (MRE) and MRct1 fibrosis classification (historical records) and to assess LIVERFASt performance for MR steatosis assessment in an United States adult miscellaneous population with available (historical) MR intracellular fat fraction assessment (ICFF) from a single tertiary US clinic.

DETAILED DESCRIPTION:
1. To assess the correlation and the strength of concordance of LIVERFASt for staging important liver lesions of fibrosis and steatosis against MR liver assessment of clinically significant (≥F2 stage), advanced fibrosis (≥F3 stage) and cirrhosis (F4 stage) (MRE, ct1) and steatosis (MR) in a SLD (MASLD, MetALD) adult US population.
2. To assess the diagnostic performance [AUROC (95%CI)] of LIVERFASt for diagnosing important liver lesions of fibrosis, steatosis taking MR-based methods as surrogate gold-standard (MRE for fibrosis assessment and MR for steatosis quantification).

ELIGIBILITY:
Inclusion Criteria:

* SLD with MASLD or MetALD Adult patients with:

  * available historical report of MRE and LIVERFASt test
  * at least fibrosis scoring available (steatosis and necro-inflammation imaging reports are requested equally when available).
* Other imaging modality reports ie. MRI, ARFI, ct1, SWE and Fibroscan can be included when available

Exclusion Criteria:

* Participants identified as having risk factors for false positive/negative results for Liverfast (severe intravascular hemolysis-if condition is known-, acute hepatitis or severe cytolysis with ≥ 600 ALT values)
* Other comorbidities not compatible with the diagnosis of MASLD or MetALD

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • The expected number of subjects is around N=100 adult patients with Steatotic Liver Disease (MASLD or MetALD) with either paired MRE historical report and LIVERFASt or MR and LIVERFASt.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical correlation evaluation of the LIVERFAStTM Test for diagnosing important liver lesions of fibrosis and steatosis against Magnetic Resonance Elastography for Liver Fibrosis and MR-based assessment of steatosis, in adult US population. | 6 months
  1/ Two-class concordance rate (kappa, p value) between MRE and LIVERFASt fibrosis test for each of the fibrosis endpoints (≥F2, ≥F3, F4)
Clinical correlation evaluation of the LIVERFAStTM Test for diagnosing important liver lesions of fibrosis and steatosis against Magnetic Resonance Elastography for Liver Fibrosis and MR-based assessment of steatosis, in adult US population. | 6 months
  2/ AUROCs (95%CI) for fibrosis endpoints (≥F2, ≥F3, F4) and steatosis endpoints (≥S1, ≥S2 and S3) against surrogate gold-standard, MRE and MR-PDFF, respectively

SECONDARY OUTCOMES:
Clinical correlation evaluation of the LIVERFAStTM Test for diagnosing important liver lesions of fibrosis and steatosis against Magnetic Resonance Elastography for Liver Fibrosis and MR-based assessment of steatosis, in adult US population. | 6 months
  3/ Discordance analysis using independent clinical criteria (e.g. biopsy, other circulating or imaging NITs,)

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Gastroenterology & Surgery Associates, Lady Lake, Florida, United States

REFERENCES:
- See also: Related Info — https://fibronostics.com